CLINICAL TRIAL: NCT02075606
Title: A Phase IV, Multicentre, Open Label, Single Group Exploratory Study to Assess the Clinical Value of Enumeration of Circulating Tumour Cells (CTCs) to Predict Clinical Symptomatic Response and Progression Free Survival in Patients Receiving Deep Subcutaneous Administrations of Somatuline® (Lanreotide) Autogel® to Treat the Symptoms of Functioning Midgut NeuroEndocrine Tumours (NET)
Brief Title: Circulating Tumour Cells in Somatuline Autogel Treated NeuroEndocrine Tumours Patients
Acronym: CALM-NET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A-97-52030-270; 2013-002194-22 (EudraCT Number)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-02

CONDITIONS: NeuroEndocrine Tumours
Keywords: NET; Symptomatic response; Functioning NeuroEndocrine Tumours; midgut region
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Somatuline Autogel® (Experimental): Somatuline Autogel® to treat Functioning Midgut NeuroEndocrine Tumours (NET)
  Interventions: Drug: lanreotide acetate

INTERVENTIONS:
Drug: lanreotide acetate — Somatuline Autogel injection 120mg for first 3 months then 120, 90 or 60 mg administered via the deep subcutaneous route every 28 days

SUMMARY:
Circulating tumour cells (CTCs) are detectable in the blood in around 50% of patients with functioning NeuroEndocrine Tumours (NET) arising in the midgut area (tumours which are secreting hormones and are located in the area in the middle of the digestive system) and their presence usually means that the prognosis for the patient is poor. CTCs have also been shown to be valuable as predictive markers following treatment and there is increasing interest in using CTCs as 'liquid biopsies' that can help to inform treatment decisions. CTC analysis has the benefit of being relatively non- invasive and quick compared with a conventional CT scan and is therefore an attractive method of monitoring the tumour throughout the treatment period.

The purpose of this study is to assess the clinical value that enumeration will have in predicting the clinical symptomatic response and progression free survival in patients receiving Somatuline Autogel for functioning midgut NETs over a one year period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* Patients (either sex) must be 18 years or older.
* Patients must be suffering from symptoms of diarrhoea and/or flushing at the time of study enrolment.
* Patients must have a documented diagnosis of a functioning midgut NET.
* In order to avoid patients with rapidly progressing tumours, only patients with well or moderately differentiated tumours and with a Ki67 proliferation index of <20% will be recruited.
* The clinically appropriate treatment for the patient must be therapy with a somatostatin analogue.
* Patients must have had either a positive somatostatin receptor scintigraphy result or a positive 68Gallium-DOTATATE PET imaging result.

Exclusion Criteria:

* If the patient is at risk of pregnancy or is breast feeding, unless treatment with Somatuline Autogel is clearly needed (as determined by the clinician).
* The patient is, in the opinion of the investigator, unable to comply fully with the protocol and the study instructions, or present any concomitant condition which could compromise the objectives of the study and/or preclude the protocol-defined procedures (e.g. severe medical conditions, brain metastases, psychiatric disorders, active or uncontrolled infection, known pituitary disease).
* The patient has been treated with any other unlicensed drug within the last 30 days before study entry or will require a concurrent treatment with any other experimental drugs or treatments.
* The patient has been treated with a somatostatin analogue prior to study entry, unless a washout period of at least 2 weeks for subcutaneous octreotide, or at least 6 weeks for a single dose of long acting somatostatin analogue has occurred.
* The patient has received interferon, chemotherapy, chemoembolisation or radionuclide therapy within 3 months prior to study entry.
* The patient has a history of hypersensitivity to drugs with a similar chemical structure.
* Females of childbearing potential must be using oral, double barrier or injectable contraception. Non childbearing potential is defined as being post-menopause for at least 1 year, surgical sterilisation or hysterectomy at least three months before the start of the study.
* The patient has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hickling, MD, Study Director — Ipsen
Locations (14):
- United Kingdom (14):
  - Basingstoke & North Hampshire Hospital, Basingstoke
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital Wales, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - University Hospital Aintree, Liverpool
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Royal Free Hospital, London
  - Maidstone Hospital, Maidstone
  - The Christie Hospital, Manchester
  - Norfolk & Norwich Hospital, Norwich
  - Royal Hallamshire Hospital, Sheffield
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Meyer T, Caplin M, Khan MS, Toumpanakis C, Shetty S, Ramage JK, Houchard A, Higgs K, Shah T. Circulating tumour cells and tumour biomarkers in functional midgut neuroendocrine tumours. J Neuroendocrinol. 2022 Apr;34(4):e13096. doi: 10.1111/jne.13096. Epub 2022 Feb 7. PMID 35132704
- [Derived] Childs A, Vesely C, Ensell L, Lowe H, Luong TV, Caplin ME, Toumpanakis C, Thirlwell C, Hartley JA, Meyer T. Expression of somatostatin receptors 2 and 5 in circulating tumour cells from patients with neuroendocrine tumours. Br J Cancer. 2016 Dec 6;115(12):1540-1547. doi: 10.1038/bjc.2016.377. Epub 2016 Nov 22. PMID 27875519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to this prospective, pilot, phase IV, multicentre, open-label, single-group study began on 16 May 2014. Subjects with a documented diagnosis of functioning midgut NET and who suffered from symptoms of diarrhoea and/or flushing at the time of enrolment were recruited to 11 study centres in the United Kingdom.
Pre-assignment Details: Overall, 54 subjects were screened, 50 of whom were enrolled and treated in the study.
Groups:
- Lanreotide Autogel: Subjects received deep subcutaneous injections of lanreotide Autogel for 1 year to treat the symptoms of functioning midgut NETs.
  A washout period was required for subjects receiving either subcutaneous octreotide (at least 2 weeks) or 1 injection of long-acting somatostatin analogue (at least 6 weeks) prior to treatment in the study.
  Initially subjects began treatment with a dose of lanreotide Autogel 120 milligrams (mg) every 28 days for 3 months. Thereafter, the dose administered was determined on an individual subject basis by the treating clinician. Subjects could remain on the 120 mg dose, or be titrated to either 60 mg or 90 mg lanreotide Autogel, administered every 28 days according to their symptomatic response.
Period: Overall Study
Arm/Group | Lanreotide Autogel
Started | 50
Completed | 40
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Investigator's decision | 1
Not completed — Symptom management | 1
Not completed — Increasing Symptoms | 1

BASELINE CHARACTERISTICS:
Groups:
- Lanreotide Autogel: Subjects received deep subcutaneous injections of lanreotide Autogel for 1 year to treat the symptoms of functioning midgut NETs.
  A washout period was required for subjects receiving either subcutaneous octreotide (at least 2 weeks) or 1 injection of long-acting somatostatin analogue (at least 6 weeks) prior to treatment in the study.
  Initially subjects began treatment with a dose of lanreotide Autogel 120 mg every 28 days for 3 months. Thereafter, the dose administered was determined on an individual subject basis by the treating clinician. Subjects could remain on the 120 mg dose, or be titrated to either 60 mg or 90 mg lanreotide Autogel, administered every 28 days according to their symptomatic response.
Arm/Group | Lanreotide Autogel
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years]
  years | 63.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Clinical Symptomatic Response
Description: This endpoint was assessed using 2 efficacy variables:
  * CTCs, enumerated at baseline and Weeks 5, 17, 25, 53
  * Clinical symptomatic response, assessed by the use of symptom reporting
  Subjects recorded 24-hour symptom frequency and severity for 7 days prior to first treatment (baseline), throughout the study, and up to 28 days following final drug administration. Symptoms were recorded by answering predetermined questions on the interactive voice response system (IVRS).
  Subjects were considered to have a clinical symptomatic response between baseline and last study visit if any 1 of the following criteria were fulfilled: the average number of episodes of diarrhoea decreased by at least 50%, the average number of episodes of flushing decreased by at least 50%, the mode severity of flushing decreased by at least 1 level. Clinical symptomatic response was assessed as a qualitative variable (Yes/No) and reported according to CTC presence at baseline and overall.
Time Frame: From baseline up to Week 53.
Population: Analysis was performed on the Intention-to-treat (ITT) population, defined as all enrolled subjects who received at least one injection of study medication. Only subjects with data available for analysis are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- CTC Presence at Baseline: Subjects with a baseline presence of CTCs, determined by either or both baseline CTC blood samples having a CTC enumeration >0.
  Baseline is defined as the 7 days preceding the first study treatment injection, or for subjects who required a washout period, these 7 days were during the washout period.
- No CTC Presence at Baseline: Subjects with no baseline presence of CTCs, determined by both baseline CTC blood samples having a CTC enumeration = 0.
  Baseline is defined as the 7 days preceding the first study treatment injection, or for subjects who required a washout period, these 7 days were during the washout period.
Arm/Group | CTC Presence at Baseline | No CTC Presence at Baseline | Lanreotide Autogel
Number analyzed (Participants) | 22 | 26 | 50
Percentage of Subjects
  Clinical Symptomatic Response = Yes(2) | 77.8 [54.8 to 91.0] | 95.5 [78.2 to 99.2] | 87.5 [73.9 to 94.5]
  Clinical Symptomatic Response = No(3) | 22.2 [9.0 to 45.2] | 4.5 [0.8 to 21.8] | 12.5 [5.5 to 26.1]
Statistical Analysis 1: Comparison: CTC Presence at Baseline vs No CTC Presence at Baseline; Clinical symptomatic response as dependent variable and CTC presence at baseline as explanatory variable was used to perform the logistic regression analysis; Test type: Other; p = 0.126, Regression, Logistic; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.02 to 1.65]

2. Primary Outcome: Percentage of Subjects With Time Point Responses According to Response Evaluation Criteria in Solid Tumours (RECIST) Assessments at Weeks 25 and 53
Description: Subjects underwent Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scans at baseline, Visit 8 (Week 25) and Visit 15 (Week 53). Progression was assessed by investigators using RECIST v1.1, and classified as a complete response, partial response, stable disease, progressive disease or non evaluable.
  The time point responses at Week 25 and Week 53 were analysed by CTC presence at baseline and overall. The percentage of subjects within each response category are presented. Percentages are based on the number of subjects in the concerned population with available responses.
Time Frame: Week 25 and Week 53.
Population: Analysis was performed on subjects from the ITT population, defined as all enrolled subjects who received at least one injection of study medication. Only subjects with data available for analysis are presented.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CTC Presence at Baseline | No CTC Presence at Baseline | Lanreotide Autogel
Number analyzed (Participants) | 22 | 26 | 50
percentage of subjects
  Week 25: Complete Response: number analyzed (Participants) | 11 | 12 | 23
  Week 25: Complete Response | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 24.2] | 0.0 [0.0 to 14.3]
  Week 25: Partial Response: number analyzed (Participants) | 11 | 12 | 23
  Week 25: Partial Response | 18.2 [5.1 to 47.7] | 8.3 [1.5 to 35.4] | 13.0 [4.5 to 32.1]
  Week 25: Stable Disease: number analyzed (Participants) | 11 | 12 | 23
  Week 25: Stable Disease | 72.7 [43.4 to 90.3] | 75.0 [46.8 to 91.1] | 73.9 [53.5 to 87.5]
  Week 25: Progressive Disease: number analyzed (Participants) | 11 | 12 | 23
  Week 25: Progressive Disease | 9.1 [1.6 to 37.7] | 16.7 [4.7 to 44.8] | 13.0 [4.5 to 32.1]
  Week 25: Non evaluable: number analyzed (Participants) | 11 | 12 | 23
  Week 25: Non evaluable | 0.0 [0.0 to 25.9] | 0.0 [0.0 to 24.2] | 0.0 [0.0 to 14.3]
  Week 53: Complete Response: number analyzed (Participants) | 15 | 22 | 37
  Week 53: Complete Response | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 14.9] | 0.0 [0.0 to 9.4]
  Week 53: Partial Response: number analyzed (Participants) | 15 | 22 | 37
  Week 53: Partial Response | 6.7 [1.2 to 29.8] | 4.5 [0.8 to 21.8] | 5.4 [1.5 to 17.7]
  Week 53: Stable Disease: number analyzed (Participants) | 15 | 22 | 37
  Week 53: Stable Disease | 66.7 [41.7 to 84.8] | 63.6 [43.0 to 80.3] | 64.9 [48.8 to 78.2]
  Week 53: Progressive Disease: number analyzed (Participants) | 15 | 22 | 37
  Week 53: Progressive Disease | 26.7 [10.9 to 52.0] | 31.8 [16.4 to 52.7] | 29.7 [17.5 to 45.8]
  Week 53: Non evaluable: number analyzed (Participants) | 15 | 22 | 37
  Week 53: Non evaluable | 0.0 [0.0 to 20.4] | 0.0 [0.0 to 14.9] | 0.0 [0.0 to 9.4]

3. Secondary Outcome: Mean Change From Baseline in Number of Episodes of Diarrhoea and Flushing
Description: The effect of lanreotide Autogel on the symptoms of diarrhoea and flushing in subjects was assessed through subject reporting of symptoms every 24-hours for the 7 days prior to treatment (baseline), for the first 16 weeks and on days 11 to 17 after each subsequent injection interval. After the final study drug injection at Week 49, subjects provided 24-hour symptom frequency on days 11 to 28 (up to Week 53). Symptom frequency was recorded by answering predetermined questions on the IVRS.
  Mean change from baseline in frequency (number of episodes) of diarrhoea and flushing are described at Visit 2 (average number of episodes in Week 1) and at Visit 14 (average number of episodes over days 11 to 17 after Week 49 injection and over days 11 to 28 after Week 49 injection) by CTC presence at baseline and overall. A negative change indicates an improvement in symptoms from baseline.
Time Frame: From baseline up to Week 53.
Population: Analysis was performed on the ITT population, defined as all enrolled subjects who received at least one injection of study medication. Only subjects with data available for analysis at each time point are reported.
Measure: Mean (95% Confidence Interval); unit: number of episodes
Groups:
- Missing CTC Status at Baseline: Subjects whose CTC status at baseline could not be evaluated as both CTC blood samples were missing. Baseline is defined as the 7 days preceding the first study treatment injection, or for subjects who required a washout period, these 7 days were during the washout period.
Arm/Group | CTC Presence at Baseline | No CTC Presence at Baseline | Missing CTC Status at Baseline | Lanreotide Autogel
Number analyzed (Participants) | 22 | 26 | 2 | 50
number of episodes
  Diarrhoea: Visit 2 (daily): number analyzed (Participants) | 22 | 25 | 2 | 49
  Diarrhoea: Visit 2 (daily) | -0.66 [-1.68 to 0.36] | -0.27 [-0.73 to 0.20] | 0.38 [-11.18 to 11.93] | -0.42 [-0.92 to 0.08]
  Diarrhoea: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  Diarrhoea: Visit 14 (days 11-17) | -1.91 [-3.24 to 0.57] | -0.64 [-1.16 to -0.11] |  | -1.18 [-1.83 to -0.54]
  Diarrhoea: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  Diarrhoea: Visit 14 (days 11-28) | -2.15 [-3.49 to -0.82] | -0.63 [-1.19 to -0.08] |  | -1.30 [-1.98 to -0.63]
  Flushing: Visit 2 (daily): number analyzed (Participants) | 22 | 25 | 2 | 49
  Flushing: Visit 2 (daily) | -1.76 [-3.41 to -0.11] | -1.25 [-2.02 to -0.48] | 0.00 [0.00 to 0.00] | -1.43 [-2.24 to -0.62]
  Flushing: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  Flushing: Visit 14 (days 11-17) | -3.37 [-5.76 to -0.98] | -2.51 [-3.68 to -1.33] |  | -2.88 [-4.05 to -1.71]
  Flushing: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  Flushing: Visit 14 (days 11-28) | -3.49 [-6.00 to -0.99] | -2.23 [-3.34 to -1.13] |  | -2.79 [-3.99 to -1.58]

4. Secondary Outcome: Mode Symptom Severity of Episodes of Flushing
Description: The effect of lanreotide Autogel on the mode severity of flushing was assessed through subject reporting of symptoms every 24-hours for the 7 days prior to treatment (baseline), for the first 16 weeks and on days 11 to 17 after each subsequent injection interval until Week 49. After the final study drug injection at Week 49, subjects provided 24-hour symptom severity on days 11 to 28 (up to Week 53). Symptom severity was recorded by answering predetermined questions on the IVRS using a three-point system (mild, moderate or severe). The mode (most frequent) intensity of flushing are reported at baseline and at Visit 14 (average number of episodes over days 11 to 17 after Week 49 injection and over days 11 to 28 after Week 49 injection). Percentages of subjects in each severity category are based on the number of subjects in the analysis set with available responses. Data is presented according to CTC presence at baseline and overall.
Time Frame: From baseline up to Week 53.
Population: Analysis was performed on the ITT population, defined as all enrolled subjects who received at least one injection of study medication. Only subjects with data available for analysis are presented.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CTC Presence at Baseline | No CTC Presence at Baseline | Missing CTC Status at Baseline | Lanreotide Autogel
Number analyzed (Participants) | 22 | 26 | 2 | 50
percentage of subjects
  No flushing: Baseline | 22.7 [10.1 to 43.4] | 0.0 [0.0 to 12.9] | 100 [34.2 to 100] | 14.0 [7.0 to 26.2]
  Mild: Baseline | 27.3 [13.2 to 48.2] | 50.0 [32.1 to 67.9] | 0.0 [0.0 to 65.8] | 38.0 [25.9 to 51.8]
  Moderate: Baseline | 45.5 [26.9 to 65.3] | 50.0 [32.1 to 67.9] | 0.0 [0.0 to 65.8] | 46.0 [33.0 to 59.6]
  Severe: Baseline | 4.5 [0.8 to 21.8] | 0.0 [0.0 to 12.9] | 0.0 [0.0 to 65.8] | 2.0 [0.4 to 10.5]
  No flushing: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  No flushing: Visit 14 (days 11-17) | 37.5 [18.5 to 61.4] | 28.6 [13.8 to 50.0] |  | 32.4 [19.6 to 48.5]
  Mild: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  Mild: Visit 14 (days 11-17) | 43.8 [23.1 to 66.8] | 47.6 [28.3 to 67.6] |  | 45.9 [31.0 to 61.6]
  Moderate: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  Moderate: Visit 14 (days 11-17) | 18.8 [6.6 to 43.0] | 23.8 [10.6 to 45.1] |  | 21.6 [11.4 to 37.2]
  Severe: Visit 14 (days 11-17): number analyzed (Participants) | 16 | 21 | 0 | 37
  Severe: Visit 14 (days 11-17) | 0.0 [0.0 to 19.4] | 0.0 [0.0 to 15.5] |  | 0.0 [0.0 to 9.4]
  No flushing: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  No flushing: Visit 14 (days 11-28) | 13.3 [3.7 to 37.9] | 31.6 [15.4 to 54.0] |  | 23.5 [12.4 to 40.0]
  Mild: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  Mild: Visit 14 (days 11-28) | 60.0 [35.7 to 80.2] | 52.6 [31.7 to 72.7] |  | 55.9 [39.5 to 71.1]
  Moderate: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  Moderate: Visit 14 (days 11-28) | 26.7 [10.9 to 52.0] | 10.5 [2.9 to 31.4] |  | 17.6 [8.3 to 33.5]
  Severe: Visit 14 (days 11-28): number analyzed (Participants) | 15 | 19 | 0 | 34
  Severe: Visit 14 (days 11-28) | 0.0 [0.0 to 20.4] | 5.3 [0.9 to 24.6] |  | 2.9 [0.5 to 14.9]

5. Secondary Outcome: Quality of Life (QoL) Questionnaire: European Organisation for Research and Treatment of Cancer (EORTC) QoL Questionnaire (QLQ)-C30
Description: The effect of lanreotide Autogel treatment on QoL was assessed using the EORTC QLQ-C30 at baseline, Weeks 13 (Visit 5), 25 (Visit 8) and 53 (Visit 15/end of study). The 30 item scale is divided into 9 multi item scales (including 5 functional scales, 1 global health status/QoL scale and 3 general symptom scales) and 6 single items. Possible answers to the first 28 items (all items except the 2 concerning global quality of life) go from 1 (Not at all) to 4 (Very much). The answers for the 2 last questions (Q29- 30) go from 1 (Very poor) to 7 (Excellent). All of the scales and single-item measures range in score from 0 to 100. For multi-item scales, the raw score will be calculated by the addition of item responses divided by the number of items. Higher scores for global health and functional domains indicate a better QoL, while higher symptom scores indicate worse symptoms.
  The mean change from baseline at each time point is reported for each of the category subscores.
Time Frame: From baseline up to Week 53.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lanreotide Autogel
Number analyzed (Participants) | 50
Units on a scale
  Physical functioning: Visit 5: number analyzed (Participants) | 39
  Physical functioning: Visit 5 | 1.2 (17.9)
  Physical functioning: Visit 8: number analyzed (Participants) | 36
  Physical functioning: Visit 8 | 2.0 (17.6)
  Physical functioning: End of study: number analyzed (Participants) | 36
  Physical functioning: End of study | 1.9 (21.7)
  Role functioning: Visit 5: number analyzed (Participants) | 39
  Role functioning: Visit 5 | 1.3 (30.9)
  Role functioning: Visit 8: number analyzed (Participants) | 36
  Role functioning: Visit 8 | 3.2 (32.1)
  Role functioning: End of study: number analyzed (Participants) | 36
  Role functioning: End of study | -1.4 (33.7)
  Emotional functioning: Visit 5: number analyzed (Participants) | 36
  Emotional functioning: Visit 5 | 6.1 (24.8)
  Emotional functioning: Visit 8: number analyzed (Participants) | 34
  Emotional functioning: Visit 8 | 4.3 (18.3)
  Emotional functioning: End of study: number analyzed (Participants) | 35
  Emotional functioning: End of study | 1.1 (23.0)
  Cognitive functioning: Visit 5: number analyzed (Participants) | 36
  Cognitive functioning: Visit 5 | -0.9 (19.9)
  Cognitive functioning: Visit 8: number analyzed (Participants) | 34
  Cognitive functioning: Visit 8 | 1.5 (15.6)
  Cognitive functioning: End of study: number analyzed (Participants) | 35
  Cognitive functioning: End of study | -2.4 (19.9)
  Social functioning: Visit 5: number analyzed (Participants) | 35
  Social functioning: Visit 5 | 10.0 (26.9)
  Social functioning: Visit 8: number analyzed (Participants) | 33
  Social functioning: Visit 8 | 4.5 (30.1)
  Social functioning: End of study: number analyzed (Participants) | 34
  Social functioning: End of study | 3.9 (27.8)
  Global QoL: Visit 5: number analyzed (Participants) | 36
  Global QoL: Visit 5 | 12.5 (26.4)
  Global QoL: Visit 8: number analyzed (Participants) | 34
  Global QoL: Visit 8 | 7.4 (24.3)
  Global QoL: End of study: number analyzed (Participants) | 35
  Global QoL: End of study | 4.3 (22.8)
  Fatigue: Visit 5: number analyzed (Participants) | 39
  Fatigue: Visit 5 | -4.4 (26.7)
  Fatigue: Visit 8: number analyzed (Participants) | 36
  Fatigue: Visit 8 | -6.3 (21.2)
  Fatigue: End of study: number analyzed (Participants) | 36
  Fatigue: End of study | -4.2 (25.6)
  Nausea and vomiting: Visit 5: number analyzed (Participants) | 40
  Nausea and vomiting: Visit 5 | -4.2 (20.9)
  Nausea and vomiting: Visit 8: number analyzed (Participants) | 37
  Nausea and vomiting: Visit 8 | -1.4 (20.9)
  Nausea and vomiting: End of study: number analyzed (Participants) | 37
  Nausea and vomiting: End of study | -0.9 (29.1)
  Pain: Visit 5: number analyzed (Participants) | 40
  Pain: Visit 5 | -7.9 (32.5)
  Pain: Visit 8: number analyzed (Participants) | 37
  Pain: Visit 8 | -2.3 (30.2)
  Pain: End of study: number analyzed (Participants) | 37
  Pain: End of study | 1.8 (30.6)
  Dyspnoea: Visit 5: number analyzed (Participants) | 38
  Dyspnoea: Visit 5 | -3.5 (25.5)
  Dyspnoea: Visit 8: number analyzed (Participants) | 35
  Dyspnoea: Visit 8 | 1.0 (20.6)
  Dyspnoea: End of study: number analyzed (Participants) | 35
  Dyspnoea: End of study | -4.8 (30.4)
  Insomnia: Visit 5: number analyzed (Participants) | 37
  Insomnia: Visit 5 | -6.3 (27.0)
  Insomnia: Visit 8: number analyzed (Participants) | 35
  Insomnia: Visit 8 | -5.7 (22.1)
  Insomnia: End of study: number analyzed (Participants) | 34
  Insomnia: End of study | -2.9 (37.0)
  Appetite loss: Visit 5: number analyzed (Participants) | 34
  Appetite loss: Visit 5 | -0.9 (37.1)
  Appetite loss: Visit 8: number analyzed (Participants) | 36
  Appetite loss: Visit 8 | -6.5 (36.4)
  Appetite loss: End of study: number analyzed (Participants) | 36
  Appetite loss: End of study | -0.0 (34.7)
  Constipation: Visit 5: number analyzed (Participants) | 36
  Constipation: Visit 5 | 1.9 (19.4)
  Constipation: Visit 8: number analyzed (Participants) | 33
  Constipation: Visit 8 | -1.0 (13.1)
  Constipation: End of study: number analyzed (Participants) | 35
  Constipation: End of study | 1.9 (13.9)
  Diarrhoea: Visit 5: number analyzed (Participants) | 36
  Diarrhoea: Visit 5 | -18.5 (33.3)
  Diarrhoea: Visit 8: number analyzed (Participants) | 34
  Diarrhoea: Visit 8 | -12.7 (30.7)
  Diarrhoea: End of study: number analyzed (Participants) | 34
  Diarrhoea: End of study | -10.8 (32.5)
  Financial difficulties: Visit 5: number analyzed (Participants) | 35
  Financial difficulties: Visit 5 | -6.7 (25.3)
  Financial difficulties: Visit 8: number analyzed (Participants) | 33
  Financial difficulties: Visit 8 | -4.0 (30.9)
  Financial difficulties: End of study: number analyzed (Participants) | 34
  Financial difficulties: End of study | -1.0 (38.0)

6. Secondary Outcome: QoL Questionnaire: EORTC QLQ-G.I.NET21
Description: The effect of lanreotide Autogel treatment on QoL was assessed using the EORTC QLQ-G.I.NET21 at baseline, Weeks 13 (Visit 5), 25 (Visit 8) and 53 (Visit 15/end of study). The QLQ-G.I.NET21 questionnaire contained 21 questions that used a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much) to evaluate 3 defined multi-item symptom scales (endocrine, gastrointestinal and treatment related side effects), 2 single item symptoms (bone/muscle pain and concern about weight loss), 2 psychosocial scales (social function and disease-related worries) and 2 other single items (sexuality and communication). Each individual subscore was transformed to range from 0 to 100. Higher scores indicate worse symptoms or more problems. The mean change from baseline at each time point is reported for each of the category subscores.
Time Frame: From baseline up to Week 53.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lanreotide Autogel
Number analyzed (Participants) | 50
Units on a scale
  Endocrine symptoms: Visit 5: number analyzed (Participants) | 39
  Endocrine symptoms: Visit 5 | -15.4 (21.6)
  Endocrine symptoms: Visit 8: number analyzed (Participants) | 37
  Endocrine symptoms: Visit 8 | -17.0 (22.9)
  Endocrine symptoms: End of study: number analyzed (Participants) | 36
  Endocrine symptoms: End of study | -16.0 (22.8)
  Gastrointestinal symptoms: Visit 5: number analyzed (Participants) | 39
  Gastrointestinal symptoms: Visit 5 | 2.1 (16.9)
  Gastrointestinal symptoms: Visit 8: number analyzed (Participants) | 37
  Gastrointestinal symptoms: Visit 8 | 1.2 (15.6)
  Gastrointestinal symptoms: End of study: number analyzed (Participants) | 36
  Gastrointestinal symptoms: End of study | 1.0 (16.7)
  Treatment symptoms: Visit 5: number analyzed (Participants) | 9
  Treatment symptoms: Visit 5 | 1.2 (15.2)
  Treatment symptoms: Visit 8: number analyzed (Participants) | 8
  Treatment symptoms: Visit 8 | 7.6 (8.9)
  Treatment symptoms: End of study: number analyzed (Participants) | 6
  Treatment symptoms: End of study | 12.0 (12.4)
  Social function: Visit 5: number analyzed (Participants) | 39
  Social function: Visit 5 | -11.3 (26.6)
  Social function: Visit 8: number analyzed (Participants) | 37
  Social function: Visit 8 | -6.5 (29.3)
  Social function: End of study: number analyzed (Participants) | 36
  Social function: End of study | -4.5 (24.1)
  Disease related worries: Visit 5: number analyzed (Participants) | 39
  Disease related worries: Visit 5 | -14.1 (25.2)
  Disease related worries: Visit 8: number analyzed (Participants) | 37
  Disease related worries: Visit 8 | -15.9 (33.8)
  Disease related worries: End of study: number analyzed (Participants) | 36
  Disease related worries: End of study | -12.2 (36.3)
  Muscle/Bone pain: Visit 5: number analyzed (Participants) | 38
  Muscle/Bone pain: Visit 5 | -7.9 (36.7)
  Muscle/Bone pain: Visit 8: number analyzed (Participants) | 36
  Muscle/Bone pain: Visit 8 | -6.5 (31.7)
  Muscle/Bone pain: End of study: number analyzed (Participants) | 34
  Muscle/Bone pain: End of study | -11.8 (39.3)
  Sexual function: Visit 5: number analyzed (Participants) | 18
  Sexual function: Visit 5 | -5.6 (34.8)
  Sexual function: Visit 8: number analyzed (Participants) | 15
  Sexual function: Visit 8 | -8.9 (34.4)
  Sexual function: End of study: number analyzed (Participants) | 15
  Sexual function: End of study | -13.3 (27.6)
  Information/communication function: Visit 5: number analyzed (Participants) | 39
  Information/communication function: Visit 5 | -8.5 (26.2)
  Information/communication function: Visit 8: number analyzed (Participants) | 36
  Information/communication function: Visit 8 | -3.7 (31.7)
  Information/communication function: End of study: number analyzed (Participants) | 36
  Information/communication function: End of study | -5.6 (25.8)
  Body image: Visit 5: number analyzed (Participants) | 36
  Body image: Visit 5 | 0.9 (41.0)
  Body image: Visit 8: number analyzed (Participants) | 35
  Body image: Visit 8 | 1.9 (41.2)
  Body image: End of study: number analyzed (Participants) | 35
  Body image: End of study | -1.0 (35.8)

7. Secondary Outcome: Percentage of Subjects Alive and Progression Free at One Year
Description: Subjects underwent CT or MRI scans at baseline and Week 53. Progression was assessed by investigators using RECIST v1.1. The best overall response to study treatment is the highest time point response achieved by the subject and was assessed as a complete response, partial response, stable disease, progressive disease or non evaluable. For analysis of PFS, event dates were assigned to the first time that progressive disease was noted or the date of death. In case of progressive disease followed by death, the first event was considered in the analysis. Censoring dates were defined in subjects with no progressive disease or death before end of study.
  At one year (end of study), the mean percentage of subjects who were alive and progression free, as calculated using the Kaplan-Meier method, is reported by CTC presence and overall.
Time Frame: From baseline up to Week 53.
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CTC Presence at Baseline | No CTC Presence at Baseline | Lanreotide Autogel
Number analyzed (Participants) | 22 | 26 | 50
percentage of subjects | 69.00 [40.3 to 85.94] | 67.75 [43.42 to 83.39] | 66.43 [48.77 to 79.22]

ADVERSE EVENTS:
Time Frame: From baseline to Week 53 (approximately 1 year).
Description: Treatment emergent adverse events are reported and defined as any adverse event that occurred from the first study drug injection until 28 days after the last study drug injection.
Arm/Group | Lanreotide Autogel
All-Cause Mortality (participants affected / at risk) | 3/50
Serious Adverse Events (participants affected / at risk) | 12/50
Other Adverse Events (participants affected / at risk) | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=50)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Biopsy lymph gland (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Campylobacter test positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (N=50)
Palpitations (Cardiac disorders) | 5 (6)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 16 (20)
Abdominal pain upper (Gastrointestinal disorders) | 11 (14)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 24 (29)
Flatulence (Gastrointestinal disorders) | 5 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (16)
Vomiting (Gastrointestinal disorders) | 7 (13)
Chest pain (General disorders) | 3 (5)
Fatigue (General disorders) | 16 (19)
Injection site mass (General disorders) | 5 (6)
Hepatic pain (Hepatobiliary disorders) | 3 (3)
Ear infection (Infections and infestations) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 7 (8)
Nasopharyngitis (Infections and infestations) | 6 (7)
Weight decreased (Investigations) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Dizziness (Nervous system disorders) | 12 (16)
Headache (Nervous system disorders) | 11 (25)
Sciatica (Nervous system disorders) | 3 (4)
Tremor (Nervous system disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Flushing (Vascular disorders) | 7 (9)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02075606/SAP_000.pdf
  • Study Protocol (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT02075606/Prot_001.pdf